CLINICAL TRIAL: NCT03870256
Title: The Effect of Oral Tranexamic Acid Plus, Sublingual Misoprostol in the Management of Atonic Postpartum Hemorrhage (PPH) After Vaginal Delivery: a Randomized Controlled Trial
Brief Title: Oral Tranexamic Acid Plus Sublingual Misoprostol in Atonic Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aswu/200/19
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Post Partum Hemorrhage
Keywords: Postpartum Hemorrhage; vaginal delivery; tranexamic acid; misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; carbetocin

STUDY DESIGN:
Intervention Model Description: This study was a prospective double-blind randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was a prospective double-blind randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TA plus misoprostol (Active Comparator): Patient receive 600mic gm sublingual misoprostol plus oral tranexamic acid 1 gm
  Interventions: Drug: misoprostol; Drug: TA
- Carbetocin (Active Comparator): Patient receives 100 mic gm carbetocin IV
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: misoprostol — Patient receive 600mic gm sublingual misoprostol
  Other Names: Active comparator
  Arms: TA plus misoprostol
Drug: Carbetocin — Patient receive 100 mic gm carbetocin IV
  Other Names: Active Comparator
  Arms: Carbetocin
Drug: TA — The patient receives 1gm oral tranexamic acid
  Other Names: Active Comparator
  Arms: TA plus misoprostol

SUMMARY:
The aim of the study is to evaluate the effect of oral tranexamic acid plus, sublingual misoprostol in the management of atonic postpartum hemorrhage (PPH) after vaginal delivery

DETAILED DESCRIPTION:
Uterine atony is the main cause of PPH; therefore, active management of the third stage of labor has emerged as a most actual tool in its prevention. The previous study in Egypt recorded that 88% of deaths from PPH occur within 4 h of delivery. Tranexamic acid (TA) is an antifibrinolytic agent that blocks the lysine-binding site of plasminogen to fibrin. Accordingly, clot breaks down, fibrinolysis is inhibited, and excessive bleeding is reduced. In previous studies, its safety has been confirmed for use in non-pregnant women, with no thromboembolic complications. TA is an inexpensive, widely available medicine that has been shown to reduce bleeding in surgery and reduce the risk of death in bleeding trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* All participants had PPH defined as vaginal bleeding>500 ml after vaginal delivery and uterine atony confirmed by abdominal palpation.

Exclusion Criteria:

* were gestational age<37 weeks,
* genital tract trauma,
* coagulation defect,
* women with hypertension, preeclampsia, cardiac, renal or liver diseases, epilepsy
* known hypersensitivity to carbetocin or oxytocin.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All participants had PPH defined as vaginal bleeding>500 ml after vaginal delivery and uterine atony confirmed by abdominal palpation.
Enrollment: 135 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
the amount of blood loss | 6 hours post delivery
  the amount of blood loss by gm calculated by gravimetric methods

SECONDARY OUTCOMES:
number of patients loss more than 1000 ml blood | 24 hours post delivery
  calculate number of patients loss more than 1000 ml blood
need of uterotonics | 24 hours post delivery
  number of patients need of uterotonics

CONTACTS AND LOCATIONS:
Overall Officials: hany f allam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- AswanUH, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No